CLINICAL TRIAL: NCT03907384
Title: The Effects of Mat Pilates Training on Vascular Function in Obese Premenopausal Women With Elevated Blood Pressure
Brief Title: Mat Pilates and Vascular Function in Obese Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marymount University (Other)
Collaborators: Busan University (Unknown); Texas Tech University (Other); University of Isfahan (Other)
Responsible Party: Principal Investigator, Alexei Wong, Assistant Professor, Marymount University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1342019
Record Dates: First submitted 2019-03-26; First posted 2019-04-09 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Obese; Elevated Blood Pressure
MeSH Terms: conditions — Obesity; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mat Pilates training (Experimental): The MPT group participated in 3-one hour supervised training sessions per week for 12 weeks. All MP sessions were performed in nonconsecutive days. The MP sessions were divided into the following stages: initial warm up and stretching (10 min), general conditioning consisting of MP exercises (40 min) and stretching and cooling down (10 min). The participants performed 12 basic MP exercises (one set of 6-10 repetitions was performed per exercise). Breathing, a core principle of MP, was performed by forced but controlled inspirations and exhalations, while relaxing and contracting the abdomen, respectively. All sessions were supervised by a certified MP instructor.
  Interventions: Behavioral: Mat Pilates training
- Control (No Intervention): Participants in the non-exercising control group did not participate in a supervised exercise program and visited the laboratory at the same frequency as participants in the swim intervention and underwent recreational activities such as board games

INTERVENTIONS:
Behavioral: Mat Pilates training — This group completed 12-weeks of training
  Arms: Mat Pilates training

SUMMARY:
Obesity is associated with progressive decreases in arterial health and function. It is crucial to prevent or reduce the negative effects of aging on the vasculature by implementing appropriate lifestyle interventions, such as exercise training. We examined the effects of a Mat Pilates training (MPT) regimen on arterial stiffness (pulse wave velocity, PWV), blood pressure (BP), wave reflection (AIx) and endothelial function in obese premenopausal women with elevated BP.

DETAILED DESCRIPTION:
Using a parallel experimental design, participants were randomly assigned to either MPT (n=14) or non-exercising control group (n=14) for 12 weeks. Participant in the MPT group trained 3 days/week . Participants' brachial to ankle PWV (baPWV), systolic and diastolic BP, AIx, plasma NO levels were measured at baseline and after 20 weeks of their assigned intervention.

ELIGIBILITY:
Inclusion Criteria:

* body mass index 30-40 kg/m2
* <1 h of regular exercise per week in the previous year
* systolic/diastolic BP: 120-129mm Hg systolic BP and ˂ 80 mm Hg for diastolic BP
* Nonsmokers

Exclusion Criteria:

* body mass index ˂30 and ≥40 kg/m2
* chronic diseases
* taking oral contraceptives
* pregnancy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Arterial Stiffness | 12 weeks
  via Pulse Wave Velocity

SECONDARY OUTCOMES:
Systolic and Diastolic Blood Pressure | 12 weeks
  Automatic BP monitor
Pressure Wave Reflection | 12 weeks
  via Augmentation Index
Endothelial Function | 12 weeks
  via plasma nitric oxide

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nebraska, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Wong A, Figueroa A, Fischer SM, Bagheri R, Park SY. The Effects of Mat Pilates Training on Vascular Function and Body Fatness in Obese Young Women With Elevated Blood Pressure. Am J Hypertens. 2020 May 21;33(6):563-569. doi: 10.1093/ajh/hpaa026. PMID 32236522